CLINICAL TRIAL: NCT04610788
Title: Understanding Right Ventricular Heart Failure in Scleroderma and Idiopathic Pulmonary Arterial Hypertension
Brief Title: Cardiac Assessment by PV Loop in IPAH and Scleroderma PAH
Acronym: CALIPSO
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00049022; R01HL114910-06 (NIH)
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Scleroderma; Pulmonary Artery Hypertension
MeSH Terms: conditions — Scleroderma, Diffuse; Familial Primary Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Cardiac biopsy, 4 teaspoons of blood
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- SSc-PAH Group: Scleroderma patients referred for a clinically indicated right heart catheterization (RHC).
- IPAH Group: Presumed/known IPAH patients referred for a clinically indicated right heart catheterization (RHC).

SUMMARY:
This observational study is being done to understand why people with scleroderma can develop pulmonary arterial hypertension (high blood pressure in the lungs, abbreviated PAH) and a weak heart muscle (heart failure). The study will also help the investigators understand why people with PAH from an unknown cause (called idiopathic PAH, or IPAH) can also develop a weakened heart muscle. The response of the right side of the heart or right ventricle (RV) to standard PAH therapy in scleroderma-associated PAH and in IPAH will be assessed. Blood and tissue samples will be collected from research participants during participants' normal standard of care procedures. People with scleroderma-associated PAH or idiopathic cause (IPAH) who need a right heart catheterization may join this study.

DETAILED DESCRIPTION:
Patients with scleroderma associated pulmonary hypertension (with or without interstitial lung disease) have a worse prognosis compared to patients with idiopathic pulmonary arterial hypertension (IPAH). The investigators have discovered through a previous protocol that patients with scleroderma associated pulmonary hypertension (SSc-PAH) have intrinsic right ventricular (RV) contractile dysfunction compared with patients with idiopathic pulmonary hypertension (IPAH) despite similar afterload imposed by the pulmonary vasculature. Patients with scleroderma or presumed/known IPAH who are clinically referred for right heart catheterization (RHC) will undergo, in addition to a clinically indicated RHC, state-of-the-art Pressure-Volume (P/V) Loop Assessment and RV biopsy for research purposes. The investigators will also do a standard pathologic assessment of the RV tissue (H&E, special staining, electron microscopy), microvascular density measurements using immunohistochemistry techniques and isolated skinned myocyte experiments. Additional experiments will include proteomics, genomics/genetics, and RV protein and microRNA expression. The investigators will compare these findings in both groups (IPAH and SSc-PAH), before and after standard treatment for 6 months, in order to fully understand the differences in how the RV adapts to pressure overload and reasons for impaired RV function in SSc-PAH as well as identifying potential therapeutic targets.

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years or older with clinically diagnosed scleroderma or presumed/known idiopathic pulmonary hypertension.

Exclusion Criteria:

* Patients found to have secondary pulmonary hypertension (PH due to left heart failure) on clinical RHC.
* Hemodynamically unstable patients (systolic blood pressure < 90mmHg, vasopressor requirement).
* Patients whom are unable to give consent for themselves.
* Patients with RV clot or septal aneurysm will be excluded.
* In order to undergo the clinical right heart catheterization procedures, pregnancy testing (urine or serum) is standard of care.
* Pregnancy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older with clinically diagnosed scleroderma or presumed/known idiopathic pulmonary hypertension.
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2019-04-15 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Right Ventricular Function as assessed by RHC | Baseline
  Assessed on the clinical RHC as normal, moderately reduced, or severely reduced.
Change in pulmonary vascular resistance | Baseline and 6months
  Assessed as improved or decreased after 6 months by comparing the change in pulmonary vascular resistance in Wood units on the clinical RHC.
Change in arterial elastance | Baseline and 6 months
  Assessed as improved or decreased after 6 months by comparing the change in arterial elastance in pressure volume (PV) loops.
Change in myofilament contractility | up to 4 years
  Assessed as Normal or Abnormal after studying the collected samples in lab. Abnormal can be either reduced or increased; i.e. hyper- or hypo-contractile.
Change in calcium sensitivity | up to 4 years
  Assessed as either increased- or decreased- sensitivity after 6 months, by studying the collected samples in lab.

SECONDARY OUTCOMES:
Number of genes expressed | up to 4 years
  Gene expression as assessed by observing presence of microRNA in the lab.
Number of proteins expressed | up to 4 years
  Protein expression as assessed by observing post-translational modification of candidate proteins in the lab.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Hassoun, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States